CLINICAL TRIAL: NCT04493970
Title: Assessment of Factors Impacting High School Students Mandatory Universal Student Instruction in Cardiopulmonary Resuscitation Appraised Learning- Is the Mandate Working? (The High School MUSICAL Study)
Brief Title: HS Students Mandatory Universal Student Instruction in CPR Appraised Learning- Is the Mandate Working?
Status: Recruiting | Type: Observational
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRF-High School Musical-0005
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Sudden Cardiac Arrest
Keywords: CPR Education; High School Students
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High School Students Survey — To assess retention, effectiveness and factors impacting comprehension of cardiopulmonary resuscitation (CPR) training among high school students.

SUMMARY:
This study will help to provide better input to state health and education departments to improve the processes for CPR education. This will also help the EP council explore the opportunities to partner with other professional societies and other stake holders that have interest in this topic. Engagement of private-public partnerships for improving overall CPR education.

DETAILED DESCRIPTION:
Schools should incorporate CPR education programs in the schools that will increase the knowledge, skills and awareness among high school children. It is important to note that, CPR training of young children, increases the self confidence, esteem, responsibility and contribution to their community.Moreover, it is clearly shown that, high school children has the required physical strength, maturity and positive attitude towards performing CPR in family members, friends and strangers in the community. Although some studies suggest benefit of periodic retraining, few studies have attempted to collectively identify contributing factors to comprehension.It is an attempt to identify national distribution of training efforts and factors implicated in comprehension among high school students.

ELIGIBILITY:
Inclusion Criteria:

* High school students completing voluntary survey

Exclusion Criteria:

* Inability to give consent
* Inability to complete survey

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: High school students to whom survey is distributed. Males and females will be enrolled if they meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
To assess retention, effectiveness and factors impacting comprehension of cardiopulmonary resuscitation (CPR) training among high school students. | 7 months
  To assess retention, effectiveness and factors impacting comprehension of cardiopulmonary resuscitation (CPR) training among high school students.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sudden Cardiac Arrest Foundation. 2017. Sudden cardiac arrest: A healthcare crisis. Retrieved from http://www.scaaware.org/about-sca
- [Background] Carragher, R., Johnson, J., & Harder, M. (2017). Factors that influence bystander CPR: A narrative review. International Journal of Current Research, 9(6), 52100- 52103
- [Background] Swor R, Khan I, Domeier R, Honeycutt L, Chu K, Compton S. CPR training and CPR performance: do CPR-trained bystanders perform CPR? Acad Emerg Med. 2006 Jun;13(6):596-601. doi: 10.1197/j.aem.2005.12.021. Epub 2006 Apr 13. PMID 16614455
- [Background] American Heart Association. I. CPR in schools. [cited 2019 November 29]; available from: http://cpr.heart.org/AHAECC/CPRAndECC/Programs/CPRInSchools/UCM_475820_ CPR-in-Schools-Legislation-Map.jsp; 2016
- [Background] Brown LE, Carroll T, Lynes C, Tripathi A, Halperin H, Dillon WC. CPR skill retention in 795 high school students following a 45-minute course with psychomotor practice. Am J Emerg Med. 2018 Jun;36(6):1110-1112. doi: 10.1016/j.ajem.2017.10.026. Epub 2017 Oct 13. No abstract available. PMID 29055618
- [Background] Cave DM, Aufderheide TP, Beeson J, Ellison A, Gregory A, Hazinski MF, Hiratzka LF, Lurie KG, Morrison LJ, Mosesso VN Jr, Nadkarni V, Potts J, Samson RA, Sayre MR, Schexnayder SM; American Heart Association Emergency Cardiovascular Care Committee; Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; Council on Cardiovascular Diseases in the Young; Council on Cardiovascular Nursing; Council on Clinical Cardiology, and Advocacy Coordinating Committee. Importance and implementation of training in cardiopulmonary resuscitation and automated external defibrillation in schools: a science advisory from the American Heart Association. Circulation. 2011 Feb 15;123(6):691-706. doi: 10.1161/CIR.0b013e31820b5328. Epub 2011 Jan 10. No abstract available. PMID 21220728
- [Background] Bernardo LM, Doyle C, Bryn S. Basic emergency lifesaving skills (BELS): a framework for teaching skills to children and adolescents. Int J Trauma Nurs. 2002 Apr-Jun;8(2):48-50. doi: 10.1067/mtn.2002.123027. No abstract available. PMID 12000907
- [Background] Parnell MM, Pearson J, Galletly DC, Larsen PD. Knowledge of and attitudes towards resuscitation in New Zealand high-school students. Emerg Med J. 2006 Dec;23(12):899-902. doi: 10.1136/emj.2006.041160. PMID 17130593
- [Background] Awwma Ma, A, Kl W, Ayl T, L Vyas, J Wilks. CPR knowledge and attitudes among high school students aged 15-16in Hong Kong. Hong Journal of Emergency Medicine Vol 22, Issue 1, 2015
- [Background] Chung CH. Extending cardiopulmonary resuscitation training to schools. Hong Kong J Emerg Med 2007;14:(3):131-3
- [Background] Oschatz E, Wunderbaldinger P, Sterz F, Holzer M, Kofler J, Slatin H, Janata K, Eisenburger P, Bankier AA, Laggner AN. Cardiopulmonary resuscitation performed by bystanders does not increase adverse effects as assessed by chest radiography. Anesth Analg. 2001 Jul;93(1):128-33. doi: 10.1097/00000539-200107000-00027. PMID 11429353
- [Background] Mejicano GC, Maki DG. Infections acquired during cardiopulmonary resuscitation: estimating the risk and defining strategies for prevention. Ann Intern Med. 1998 Nov 15;129(10):813-28. doi: 10.7326/0003-4819-129-10-199811150-00014. PMID 9841588
- [Background] Nabou L. Medico legal aspect of bystander CPR. Paper presented at the Hong Kong Resuscitation Council 2nd Annual Scientific Meeting, Hong Kong, 13 July 2013
- [Background] Uhm TH, Oh JK, Park JH, Yang SJ, Kim JH.Correlation between physical features of elementary school children and chest compression depth. Hong Kong J Emerg Med 2010;17(3):218-23